CLINICAL TRIAL: NCT00243490
Title: Prospective, Open-labeled, Clinical Trial in Compassionate Use to Evaluate the Efficacy and Safety of Photodynamic Therapy in the Treatment of Malignant Intracranial Tumors
Brief Title: Photodynamic Therapy in the Treatment of Malignant Intracranial Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The Trial could not get permit from Department of Health, Taiwan; Furthermore, no research fund could support the expensive (photosensitizer) photosan
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jui-Chang Tsai, M.D. Ph.D., National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33MD01
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Malignant Intracranial Tumors; Glioblastoma Multiforme; Anaplastic Astrocytomas; Anaplastic Oligodendrogliomas; Anaplastic Ependymoma
Keywords: Photodynamic therapy; Malignant glioma; Photosan
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Ependymoma; Glioma

INTERVENTIONS:
Procedure: Photodynamic therapy using Photosan and LumaCare™ Lamp Model LC-122M

SUMMARY:
Primary Objective:

* The primary objective is to evaluate the efficacy of photodynamic therapy in the treatment of malignant intracranial tumors.

Secondary Objective:

* The secondary objective is to evaluate the safety of photodynamic therapy in the treatment of malignant intracranial tumors.

DETAILED DESCRIPTION:
After passing Photosan® allergic test, the patients will be injected intravenously with Photosan® (2mg/kg) during 15~30 minutes, 48 hours prior to a standard craniotomy. Precautions are taken not to expose the patient in the operating room to direct room or operating light and to shield the skin of the flap during operation. Steroids are withdrawn 2-3 days prior to sensitization. After maximal resection, the surface of the tumor bed will be calculated and the generated cavity kept with a balloon containing intralipid (0.1%) or saline and/or artificial spinal fluid in it. A fiber with a spherical diffuser will be centered in the cavity and the surface irradiated with red (625~635nm) Halogen light. The dose of light irradiation depends on individual condition of the patient, usually with an energy density of 100 J/cm2 at a power density of 500 mW/cm2 to 600 mW/cm2.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital inpatients over the age of 20 years and under the age of 75 years, male or female.
2. Patients who are diagnosed as primary or recurrent malignant intracranial tumors (Grade III or Grade IV gliomas defined by the World Health Organization [WHO] classification), including anaplastic astrocytomas, anaplastic oligodendrogliomas, anaplastic ependymal tumors or glioblastoma multiforme.
3. Suitable for gross total resection on the basis of imaging studies from doctor's point of view
4. Karnofsky Performance Scale (KPS) ≥ 60 for newly diagnosed tumor
5. KPS ≥ 70 for recurrent tumor
6. Life expectancy at least 3 months
7. Not pregnant or lactating.
8. Patients willing to participate in the trial and sign written informed consent

Exclusion Criteria:

1. Subject is known, suspected or has history of intolerance or allergy to porphyrin.
2. Renal dysfunction (serum creatinine > 1.5 mg/dL)
3. PT/PTT greater than 1.5 times upper limit of normal (ULN)
4. Bilirubin and liver function tests (LFTs) greater than 2 times ULN
5. Alkaline phosphatase greater than 3 times ULN
6. γ-GT greater than 3 times ULN
7. Severe cardiac disease, e.g. angina pectoris, myocardial infarction, cardiac arrhythmia, congestive heart failure (New York Heart Association Functional Classification III and IV).
8. Febrile illness and total leukocyte count < 3,000/µL and/or platelet count < 80,000/µL.
9. Implantable electronic medical device such as a pacemaker, life-sustaining electronic medical device such as an artificial heart-lung machine, contact type electronic medical device such as an electrocardiograph, others such as an artificial middle ear, artificial inner ear, metal artificial cardiac valve and gold haemostatic clip.
10. Organ transplant.
11. History or evidence of severe illness or any other condition which would make the patient, in the opinion of the investigator unsuitable for the study.
12. Significant alcohol, drug or medication abuse as judged by the investigator.
13. History of treatment with any investigational drug within four weeks before the start of study.
14. Tumors located within the cerebellum or brainstem

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Study Completion 2009-01

PRIMARY OUTCOMES:
The addition of photodynamic therapy to standard brain tumor treatments will result in a significant prolongation of time to recurrence and survival in newly diagnosed malignant intracranial tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Jui-Chang Tsai, M.D. Ph.D., Principal Investigator — National Taiwan University College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan